CLINICAL TRIAL: NCT06170593
Title: Intralesional Injections of Triamcinolone for Acne Vulgaris
Acronym: ATM-2201
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACOM Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATM-2201
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Participants will receive injections of 1% triamcinolone into at least 1 and up to 3 facial inflammatory acne lesions. Participants will return to clinic at 24, 48, 72 hours, 7 days, and 14 days following injection for follow up assessment and photography.
  Interventions: Drug: Triamcinolone Injection

INTERVENTIONS:
Drug: Triamcinolone Injection — 0.1mL of triamcinolone 1% solution per lesion

SUMMARY:
This proof-of-concept study seeks to investigate the safety of intralesional injections of triamcinolone for acne vulgaris lesions using an Intradermal Needle Adapter.

DETAILED DESCRIPTION:
This is an open-label, prospective, single-arm study. Approximately 20 subjects will be enrolled at 1 study site.

All subjects will receive treatment with the study protocol (i.e., intralesional injection with triamcinolone) at Visit 1 (Day 1). Subjects will then attend in-clinic visits at Visit 2 (24-hours post-injection), Visit 3 (48-hours post-injection), Visit 4 (72-hours post-injection), Visit 5 (Day 7), and Visit 6 (Day 14).

Efficacy assessments (target lesion assessments, photography) and safety assessments will be conducted by the Investigator at each study visit. Subjects will conduct lesion pain assessments at each study visit as well as satisfaction assessments at each post-treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline.
* Diagnosed with facial acne vulgaris.
* At least one (1) identifiable inflammatory lesion that, in the opinion of the investigator, is amenable to intralesional injection of triamcinolone.
* Able to follow study instructions and likely to complete all required visits.
* In good general health as determined by medical history at the time of screening (Investigator discretion).
* Sign the IRB-approved informed consent form (including HIPAA authorization) prior to any study-related procedures being performed

Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding.
* Known hypersensitivity or previous allergic reaction to any constituent of triamcinolone injection.
* Active cutaneous viral infection in any treatment area at Baseline.
* Have concomitant skin disease or infection (other than acne) or presence of skin comorbidities in the areas of skin where study device will be used.
* History of poor cooperation or unreliability (Investigator discretion).
* Planning to move out of the area prior to study completion.
* Subjects who are investigational site staff members or family members of such employees.
* Exposure to any other investigational /device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Safety of intralesional triamcinolone injection | 14 days
  Adverse events and changes in concomitant medications

SECONDARY OUTCOMES:
Target Lesion Erythema | 14 days
  A 5-point scale ranging from 0 (No Erythema) to 4 (Very Severe Erythema).
Target Lesion Severity | 14 days
  A 5-point scale ranging from 0 (None) to 4 (Very Severe)
Target Lesion Improvement | 14 days
  A 7-point scale ranging from 1 (Clear; 100%) to 7 (Worse)
Target Lesion Pain | 14 days
  0-10 Visual Analog Scale
Target Lesion Injection Pain | Immediately after the injection of the first target lesion and at 5 minutes post-injection
  0-10 Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Dermatology Clinical Research, Inc, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT06170593/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT06170593/ICF_001.pdf